CLINICAL TRIAL: NCT00700141
Title: Non-Interventional Study on the Use of TachoSil® During Thyroid Surgery
Brief Title: Non-Interventional Study About Treatment of Hemorrhages in Thyroid Surgery With TachoSil®
Status: Completed | Type: Observational
Sponsor: Nycomed (Industry)
Responsible Party: Medical Responsible, Nycomed Deutschland GmbH
Other Study IDs: TC-031-DE
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Results first posted 2010-04-06 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2010-04

CONDITIONS: Hemorrhage
Keywords: Tachosil; thyroid; parathyroid; fleece-bound hemostasispathologic processes; hemorrhage; thyroid surgery
MeSH Terms: conditions — Hemorrhage; Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Considering the total number of thyroid procedures in Germany (100000 - 120000 cases per year), TachoSil® is a valuable tool to support surgical haemostasis, avoiding lymph leaks and support speech-nerve saving approaches. The aim of this study was to evaluate a patient and procedure profile where TachoSil® is most beneficial.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients undergoing total or subtotal thyroidectomy

Main Exclusion Criteria:

* Contraindications, such as hypersensitivity to the active pharmaceutical ingredient or to another ingredient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients
Sampling Method: Non-Probability Sample
Enrollment: 482 (Actual)
Dates: Start 2008-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Thomas D. Bethke, MD, MBA, Study Director — Nycomed Deutschland GmbH, 78467 Konstanz, Germany
Locations (110):
- Germany (110):
  - Nycomed Deutschland GmbH, Aschaffenburg
  - Nycomed Deutschland GmbH, Aschersleben
  - Nycomed Deutschland GmbH, Bad Berka
  - Nycomed Deutschland GmbH, Bad Salzungen
  - Nycomed Deutschland GmbH, Bad Tölz
  - Nycomed Deutschland GmbH, Baden-Baden
  - Nycomed Deutschland GmbH, Bayreuth
  - Nycomed Deutschland GmbH, Berlin
  - Nycomed Deutschland GmbH, Bielefeld
  - Nycomed Deutschland GmbH, Bischofswerda
  - Nycomed Deutschland GmbH, Bochum
  - Nycomed Deutschland GmbH, Bonn
  - Nycomed Deutschland GmbH, Bottrop
  - Nycomed Deutschland GmbH, Braunschweig
  - Nycomed Deutschland GmbH, Bruchsal
  - Nycomed Deutschland GmbH, Chemnitz
  - Nycomed Deutschland GmbH, Cologne
  - Nycomed Deutschland GmbH, Coswig
  - Nycomed Deutschland GmbH, Cottbus
  - Nycomed Deutschland GmbH, Deggendorf
  - Nycomed Deutschland GmbH, Detmold
  - Nycomed Deutschland GmbH, Dinkelsbühl
  - Nycomed Deutschland GmbH, Dortmund
  - Nycomed Deutschland GmbH, Duisburg
  - Nycomed Deutschland GmbH, Düsseldorf
  - Nycomed Deutschland GmbH, Eberswalde
  - Nycomed Deutschland GmbH, Eckernförde
  - Nycomed Deutschland GmbH, Eichsfeld
  - Nycomed Deutschland GmbH, Eisenach
  - Nycomed Deutschland GmbH, Erfurt
  - Nycomed Deutschland GmbH, Erlangen
  - Nycomed Deutschland GmbH, Essen
  - Nycomed Deutschland GmbH, Frankfurt
  - Nycomed Deutschland GmbH, Frankfurt (Oder)
  - Nycomed Deutschland GmbH, Frechen
  - Nycomed Deutschland GmbH, Freudenstadt
  - Nycomed Deutschland GmbH, Fürstenfeldbruck
  - Nycomed Deutschland GmbH, Fürth
  - Nycomed Deutschland GmbH, Gelnhausen
  - Nycomed Deutschland GmbH, Gelsenkirchen
  - Nycomed Deutschland GmbH, Gera
  - Nycomed Deutschland GmbH, Göppingen
  - Nycomed Deutschland GmbH, Görlitz
  - Nycomed Deutschland GmbH, Gummersbach
  - Nycomed Deutschland GmbH, Hagen
  - Nycomed Deutschland GmbH, Halle
  - Nycomed Deutschland GmbH, Hamburg
  - Nycomed Deutschland GmbH, Hamm
  - Nycomed Deutschland GmbH, Hanau
  - Nycomed Deutschland GmbH, Hartmannsdorf
  - Nycomed Deutschland GmbH, Hausham
  - Nycomed Deutschland GmbH, Heilbronn
  - Nycomed Deutschland GmbH, Heinsberg
  - Nycomed Deutschland GmbH, Herten
  - Nycomed Deutschland GmbH, Ibbenbueren
  - Nycomed Deutschland GmbH, Ingolstadt
  - Nycomed Deutschland GmbH, Jena
  - Nycomed Deutschland GmbH, Karlsruhe
  - Nycomed Deutschland GmbH, Kassel
  - Nycomed Deutschland GmbH, Konstanz
  - Nycomed Deutschland GmbH, Köln-Lindenthal
  - Nycomed Deutschland GmbH, Langen
  - Nycomed Deutschland GmbH, Leipzig
  - Nycomed Deutschland GmbH, Lichtenfels
  - Nycomed Deutschland GmbH, Loerrach
  - Nycomed Deutschland GmbH, Lohr a. Main
  - Nycomed Deutschland GmbH, Luckenwalde
  - Nycomed Deutschland GmbH, Lübbecke
  - Nycomed Deutschland GmbH, Lübeck
  - Nycomed Deutschland GmbH, Magdeburg
  - Nycomed Deutschland GmbH, Mainz
  - Nycomed Deutschland GmbH, Mannheim
  - Nycomed Deutschland GmbH, Marburg
  - Nycomed Deutschland GmbH, Meppen
  - Nycomed Deutschland GmbH, Mettmann
  - Nycomed Deutschland GmbH, München
  - Nycomed Deutschland GmbH, Münster
  - Nycomed Deutschland GmbH, Neu-Ulm
  - Nycomed Deutschland GmbH, Neumarkt in der Oberpfalz
  - Nycomed Deutschland GmbH, Neumünster
  - Nycomed Deutschland GmbH, Neuruppin
  - Nycomed Deutschland GmbH, Nordhausen
  - Nycomed Deutschland GmbH, Nuremberg
  - Nycomed Deutschland GmbH, Oberhausen
  - Nycomed Deutschland GmbH, Oldenburg
  - Nycomed Deutschland GmbH, Pforzheim
  - Nycomed Deutschland GmbH, Potsdam
  - Nycomed Deutschland GmbH, Prien am Chiemsee
  - Nycomed Deutschland GmbH, Radebeul
  - Nycomed Deutschland GmbH, Rathenow
  - Nycomed Deutschland GmbH, Recklinghausen
  - Nycomed Deutschland GmbH, Regensburg
  - Nycomed Deutschland GmbH, Rheda-Wiedenbrück
  - Nycomed Deutschland GmbH, Rosenheim
  - Nycomed Deutschland GmbH, Rostock
  - Nycomed Deutschland GmbH, Sangerhausen
  - Nycomed Deutschland GmbH, Schwedt
  - Nycomed Deutschland GmbH, Schweinfurth
  - Nycomed Deutschland GmbH, Singen
  - Nycomed Deutschland GmbH, Solingen
  - Nycomed Deutschland GmbH, Stuttgart
  - Nycomed Deutschland GmbH, Traunstein
  - Nycomed Deutschland GmbH, Trostberg an der Alz
  - Nycomed Deutschland GmbH, Ulm
  - Nycomed Deutschland GmbH, Weimar
  - Nycomed Deutschland GmbH, Weißenfels
  - Nycomed Deutschland GmbH, Wiesbaden
  - Nycomed Deutschland GmbH, Wipperfürth
  - Nycomed Deutschland GmbH, Wismar
  - Nycomed Deutschland GmbH, Würzburg

RESULTS

PARTICIPANT FLOW:
Groups:
- TachoSil® Application: Patients with application of at least one fleece of TachoSil® during thyroid surgery
Period: Overall Study
Arm/Group | TachoSil® Application
Started | 482
Completed | 482
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TachoSil® Application
Number analyzed (Participants) | 482
Age Continuous [Mean (Standard Deviation); unit: years] — The measured value is related to the number of 465 subjects. This number differs from the overall number of baseline participants due to non-availability of this information for 17 subjects.
  years
    between 15 and 91 years | 53.33 (14.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 343
  Male | 139
Number of Participants with the Indicated Hemorrhagic Risk Present [Number; unit: participants] — Multiple risks are possible for 184 participants (out of a total of 482 participants) who are affected by preoperative hemorrhagic risk according to surgeon assessment
  participants
    Application of medicines affecting coagulation | 96
    Hereditary coagulation disorders | 4
    Liver function disorders | 3
    Disturbance of the thrombocyte hemostasis | 9
    Other risks (M.Basedow, thyroiditis, tumor) | 47
    Hyperparathyroidism | 80
Type of surgery [Number; unit: participants] — * Enuc = Enucleation in one or both sides of the thyroid gland
  * 1-ST = Subtotal or near-total resection of one side of the thyroid gland
  * HT = Total resection of one side of the thyroid gland= hemithyroidectomy
  * 2-ST = Subtotal or near-total resection of both sides of the thyroid gland
  * HT+ST = Total resection of one side=hemithyroidectomy and subtotal or neartotal resection of the contralateral side
  * TE = Total resection of both lobes of the thyroid gland=thyroidectomy
  participants
    Enuc | 5
    1-ST | 25
    HT | 83
    2-ST | 82
    HT+ST | 70
    TE | 217

OUTCOME MEASURES:

1. Primary Outcome: Assessment of TachoSil® by the Surgeon With Respect to Handling, Utility and Satisfaction in the Operation, Documented Using 10 Point Numerical Rating Scales
Description: Handling (1= very good to 10= very poor) Satisfaction (1= very satisfied to 10= totally unsatisfied) Utility (1= very useful to 10= completely useless)
Time Frame: after surgery
Population: All 482 patients included and treated with TachoSil® [= Intention to Treat population (ITT)], missing values not imputed.
  For one patient missing information in all three scales (Handling, Utility and Satisfaction in the Operation)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TachoSil® Application
Number analyzed (Participants) | 481
Units on a scale
  Handling | 2.54 (1.52)
  Satisfaction | 2.25 (1.80)
  Utility | 2.42 (1.63)

2. Secondary Outcome: Pharmacoeconomic Benefits as Assessed by the Surgeon
Description: Question: What benefits resulted from the application of TachoSil® during this operation? (different categories to be answered with yes/no)
Time Frame: peri- and post-surgery until hospital discharge
Population: All 482 patients included and treated with TachoSil®, missing values not imputed.
  Multiple answers possible.
Measure: Number; unit: participants
Arm/Group | TachoSil® Application
Number analyzed (Participants) | 482
participants
  Nerve sparing through atraumatic procedure | 355
  Saving/Shortening of operation time | 286
  Reduced probability of postoperative complications | 277
  Reduced time in overall length of hospital stay | 83
  Saving of erythrocyte concentrates | 44
  Saving of thrombocyte concentrates | 30
  Reduced time in intensive care unit | 27
  Saving of Fresh Frozen Plasma (FFP) | 26

ADVERSE EVENTS:
Time Frame: peri- and post-surgery until hospital discharge
Arm/Group | TachoSil® Application
Serious Adverse Events (participants affected / at risk) | 0/482
Other Adverse Events (participants affected / at risk) | 0/482

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No